CLINICAL TRIAL: NCT05216445
Title: An Adapted Mindfulness-based Intervention for Stress Reduction and Psychological Well-being of University Students in Pakistan: a Pilot Randomized Trial Protocol
Brief Title: Mindfulness for Stress and Well-being in University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Science and Technology, Pakistan (Other)
Responsible Party: Principal Investigator, Anum Sarfraz, Principle Investigator, National University of Science and Technology, Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0098/Ethic/01/S3H/008/DBS
Record Dates: First submitted 2021-12-19; First posted 2022-01-31 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Stress; Well-being
Keywords: Mindfulness; stress; well-being; students

STUDY DESIGN:
Masking Description: The participants and intervention facilitator will be unaware at the time of allocation that which group they are being assigned to (sealed envelopes- a randomizing researcher different from the facilitator will generate the sequences and assign an ID(1-50) to one of the groups based on the sequence). The sealed envelopes will be given to the facilitator who will open the envelope in the interview and inform the participants about their allocated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Training (Experimental): The participants in this group will receive the training for 8 weeks, with 60 minute online weekly sessions. The first session will be for 90 minutes.
  Interventions: Behavioral: Mindfulness Training
- Wait-list Control (No Intervention): The wait-list control group will not receive any intervention. Once the study has been completed they will be offered the Mindfulness Training course.

INTERVENTIONS:
Behavioral: Mindfulness Training — The Mindfulness Training will be an 8-week course, with group-based online weekly sessions. The mindfulness training, translated and adapted in Urdu, includes 8 guided audio meditations and one introductory audio recording which gives the participants an overview and introduction of the forthcoming 8-week training (e.g what mindfulness is, some common terms used repeatedly). It also includes 8 chapters, corresponding to each week and a workbook to record home practice. The training will start with an online group session after which the participants will be emailed the 1st week's reading material (chapter 1), audio recordings (for that week), home practice (for that week). At the start of every week, the participants will be emailed the required material for that week. Online sessions will be conducted weekly. The participants will also be sent poems and/or quotations relating to the week's theme and based on the session proceedings.
  Arms: Mindfulness Training

SUMMARY:
In developing countries such as Pakistan, the challenges university students face are many-fold and there is a need for an intervention that helps build students' connection with themselves, utilizing their internal resources to deal with stresses. Mindfulness-based interventions have shown effectiveness with university students in high-income countries. The current study will be testing an adaptation for students of Pakistan of an intervention (Finding Peace in a Frantic World) which is based on principles from both Mindfulness-based cognitive therapy(MBCT) and Mindfulness-based stress reduction(MBSR). The purpose of this pilot trial is to assess the feasibility and acceptability (primary outcomes) of conducting a randomized controlled trial (RCT) of an adapted Mindfulness-based intervention with a wait-list control group for university students in Pakistan to reduce stress and enhance psychological well-being (N=50), which will inform the development of a future large-scale RCT. Keeping in view the COVID-19 lockdown and economic conditions in low-and-middle-income countries (LAMICs), an online program with a remote facilitator is deemed to be more cost-effective, approachable, practical, and de-stigmatizing for students.

DETAILED DESCRIPTION:
In LAMICs, including Pakistan young adults comprise more than half of the total population (60%) many of them enrolled in universities (12.7% of the total young adult population) emphasizes the need for psychological interventions in these educational institutes.

Considering the substantial lack of a systematic approach in the development, adaptation, and implementation of mindfulness-based interventions the investigators of this study employed the first two steps of Medical Research Council Guidelines (MRC) for the development of complex interventions. This current study represents the final phase of the project, where the feasibility and acceptability of the Adapted Mindfulness Training will be assessed through a Pilot RCT. The participants will be randomly assigned to either the Mindfulness Training group or the wait-list control group. The participants in the Mindfulness Training group will have online 8-week training, with weekly online group video-conference sessions with the facilitator. Both groups will be asked to complete questionnaires for outcome measures (mindfulness, well-being and stress), one week before the training starts and one week after the training ends. At the end of the training semi-structured interviews about the training will be conducted with participants (from the Mindfulness Training) who consent. The study will examine key methodological uncertainties (recruitment methods, recruitment rate, retention rate, randomization procedures), explore the acceptability of the adapted intervention and calculation of appropriate sample sizes and preliminary responses to the intervention in order to inform a future large-scale RCT. Acceptability here refers to the assessment of whether the university students find it appropriate and according to their needs and culture. To the investigator's knowledge, there haven't been any RCTs that studied the effectiveness of an online Mindfulness training translated in Urdu and adapted for university students in Pakistan to reduce stress and enhance well-being.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* enrolled in an undergraduate or postgraduate course in a university in Pakistan.

Exclusion Criteria:

* suffering from any current diagnosed severe mental illnesses including severe depression, anxiety, hypomania, or psychotic illness
* suffering from any severe medical illness.

The criteria will be self-reported by the students at the time of registration for the training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility- recruitment method | 3 months
  The number of participants recruited by each of the four methods used for recruiting. The four methods will be: social media and student groups, university platforms, referrals and recommendations and direct email to students.
  The barriers and facilitators in each method will evaluated by the recruiters.
Feasibility-recruitment rate | 3 months
  Recruitment rate will be assessed through the number of participants who registered, number of participants screened through eligibility criteria, number of participants who start the training.
Feasibility of videoconferencing | 3 months
  The assessment of barriers in technology including number of participants unable to attend sessions due to connectivity issues, number of participants dropped during sessions due to technical problems, number and type of problems, the number of participants seek extra time due to technical problems. The utility of zoom videoconferencing functions.
Feasibility-flexible multiple weekly online sessions | 2 months
  The assessment of difficulties in conducting a multiple group format on both Saturday and Sunday for each weekly online session.
Feasibility- eligibility criteria | 3 months
  Assessed through number of participants fulfilling the eligiblity criteria from the total number of students registered, number of ineligible participants and reasons for ineligibility.
Videoconferencing - acceptability by students | 3 months
  The acceptability of videoconferencing by students will be assessed in terms of ease of use (1=not at all, 5= very much; post-intervention survey), interference of technical problems (1=not at all, 5= very much; post-intervention survey), advantages and disadvantages, overall satisfaction (1=poor, 5=excellent; post-intervention survey), suggestions for improvement (feedback interview)
Acceptability - Attrition rates | 3 months
  The number of participants who complete the training and assessments, number of participants who withdraw and drop out, reasons for withdrawal and dropout.
Acceptability -participant attendance in weekly online sessions | 2 months
  Average number of sessions attended by participants, reasons for missing sessions
Acceptability-Home practice | 2 months
  Number of participants who submit weekly worksheets, average number of worksheets submitted by participants, the different tasks completed, time spent in home practice (post-training survey).
Acceptability of mindfulness training by students- semi-structured interview | 3 months
  The interview will explore students' overall satisfaction with the adapted MBI, their perception of any possible facilitators and barriers in taking part in the adapted MBI, any system changes experienced (including familial and community relationships), any physical/ psychological adverse effects or benefits experienced during and after the adapted MBI, the students' view about the mindfulness exercises and daily tasks used in the adapted mindfulness-based intervention, the group format, the home practice, any suggestions for improvement.
Feasibility of conducting the trial -randomization | 3 months
  The types and number of difficulties in randomization.
Acceptability of randomization | 3 months
  The number of participants who consented for randomization, number of participants who refused, number of participants who changed their group, reasons for refusal and change of group.
Feasibility of online data collection | 3 months
  The procedures of outcome measures data collection procedures, and online feedback interviews
Feasibility- outcome measures | 3 months
  Feasibility of outcome measures will be assessed through the assessment completion rates by participants.

SECONDARY OUTCOMES:
Psychological well-being Scale | baseline assessment before the delivery of intervention and after 8 weeks i.e the completion of intervention
  Psychological well-being Scale is used as a measure of psychological well-being with six categories; autonomy, environmental mastery, personal growth, positive relations with others, purpose in life and self-acceptance. It consists of 42 items rated on a Likert scale ranging from 1=strongly disagree to 4=strongly agree. Higher scores indicate higher levels of psychological wellbeing.
Five Facet Mindfulness Questionnaire | baseline assessment before the delivery of intervention and after 8 weeks i.e the completion of intervention
  Five Facet Mindfulness Questionnaire is used as a measure of dispositional mindfulness. It consists of 39 items rated on a Likert scale ranging from 1=never or very rarely true to 4=very often or always true. Higher scores indicate increase in mindfulness.
Clinical Outcomes Routine Evaluation-Outcome Measure | baseline assessment before the delivery of intervention and after 8 weeks i.e the completion of intervention
  Clinical Outcomes Routine Evaluation-Outcome Measure is used as a measure of psychological distress. It consists of 34 items rated on a Likert scale ranging from 1=not at all to 4=most of the time. Higher scores indicate higher levels of psychological distress.

CONTACTS AND LOCATIONS:
Overall Officials: Salma Siddiqui, Study Chair — National University of Science and Technology, Pakistan; Julieta Galante, Study Director — University of Cambridge, UK; Siham Sikandar, Study Director — National Institute of Health, Pakistan; Anum Sarfraz, Principal Investigator — National University of Science and Technology, Pakistan
Locations (1):
- National University of Science and Technology, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No